CLINICAL TRIAL: NCT00113009
Title: A Phase II, Multi-Center, Randomized, Double-Blind, Placebo Controlled Trial of VLTS-934 in Subjects With Intermittent Claudication Secondary to Peripheral Arterial Disease
Brief Title: Trial of VLTS-934 in Subjects With Intermittent Claudication Secondary to Peripheral Arterial Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valentis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VLTS-934-123
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2006-03

CONDITIONS: Peripheral Vascular Disease
Keywords: Peripheral arterial disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

INTERVENTIONS:
Drug: VLTS-934

SUMMARY:
This is a phase II, multicenter, randomized, double-blind, placebo-controlled trial in which subjects with intermittent claudication (IC) will be randomized to receive a single treatment of VLTS-934 (84 mL, or a total of 420 mg poloxamer 188) or placebo (84 mL saline) administered as 21 intramuscular (IM) injections of 2 mL each, bilaterally into the lower extremities during one procedure to evaluate the safety, tolerability, and potential activity of VLTS-934 as compared with a saline placebo.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, randomized, double-blind, placebo-controlled trial in which subjects with IC will be randomized to receive a single treatment of VLTS-934 (84 mL, or a total of 420 mg poloxamer 188) or placebo (84 mL saline) administered as 21 intramuscular (IM) injections of 2 mL each, bilaterally into the lower extremities during one procedure to evaluate the safety, tolerability, and potential activity of VLTS-934 as compared with a saline placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peripheral arterial disease in both legs
* History of exercise limiting symptoms

Exclusion Criteria:

* Lower limb revascularization surgery with 2 months of study entry
* Diagnosis of critical limb ischemia

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148
Dates: Start 2005-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in peak walking time (PWT) with VLTS-934 from baseline to Day 90 compared to subjects receiving saline placebo

SECONDARY OUTCOMES:
To evaluate changes in total work capacity, ankle-brachial index (ABI), claudication onset time and quality of life

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Los Angeles, California
  - Mountain View, California
  - Santa Rosa, California
  - Deerfield Beach, Florida
  - DeLand, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Sarasota, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Houma, Louisiana
  - Thibodaux, Louisiana
  - Auburn, Maine
  - Baltimore, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Flint, Michigan
  - Las Vegas, Nevada
  - Buffalo, New York
  - New York, New York
  - Asheville, North Carolina
  - Akron, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Warwick, Rhode Island
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Virgina Beach, Virginia
  - Seattle, Washington